CLINICAL TRIAL: NCT06682481
Title: Beta-Cell - Liver Interactions in Situations of Modified Beta-Cell Function: From Mice to Children
Brief Title: Beta-Cell - Liver Interactions in Situations of Modified Beta-Cell Function
Status: Recruiting | Type: Observational
Sponsor: Philippe Klee, MD-PhD (Other)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Philippe Klee, MD-PhD, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: 2024-00031
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Obesity, Childhood; Type 2 Diabetes Mellitus in Obese
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with obesity: Children with obesity followed within the pediatric endocrine and diabetes unit of the University Hospitals of Geneva, Switzerland. The investigators will do prospective measures in 50 children aged 12 to 15 years, at the time of a planned oral glucose tolerance test and again, 2 years later.
  Interventions: Other: Measurement of biomarker

INTERVENTIONS:
Other: Measurement of biomarker — Measurement of blood levels of 1,5-anhydroglucitol

SUMMARY:
The investigators will measure blood levels of 1,5-anhydroglucitol in obese children with or without type 2 diabetes and correlate them with parameters related to functional beta-cell mass and glucose metabolism. The values will be compared to those obtained in healthy volunteers. The aim of the study is to test the validity of 1,5-anhydroglucitol as a novel biomarker of beta-cell mass and function in children with obesity with or without type 2 diabetes.

DETAILED DESCRIPTION:
One-center prospective study performed in collaboration between the Pediatric Endocrine and Diabetology unit of the University Hospitals of Geneva (HUG) and Prof. Pierre Maechler, Diabetes Center of the Faculty of Medicine, University of Geneva Switzerland.

1,5-anhydroglucitol (1,5-AG), a deoxyhexose present in almost all foods and forming a stable pool in human subjects, has recently been found to be correlated with functional beta-cell mass in two different mouse models of beta-cell dysfunction leading to diabetes. The decline of this biomarker precedes the development of hyperglycemia in lean b-Phb2 -/- and obese db/db diabetic mice, where beta-cell loss occurs through two different mechanisms.

Additional studies have shown a correlation of 1,5-AG levels with risk of progression of type 1 diabetes (T1DM) in auto-antibody positive children, as well as with glycaemic control in patients with type 2 diabetes (T2DM).

The present project will analyse the correlation between functional beta-cell mass and the circulating levels of 1,5-AG in children with obesity with or without T2DM. This should contribute to the evaluation of a novel biomarker of beta-cell mass and function in T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12 to 16 years
* Obesity. Defined as a body-mass index above the 97th percentile.
* Ability to give informed consent as documented by signature

Exclusion Criteria:

* Patients with diabetes mellitus and positive autoantibodies against islets, insulin, islet antigen 2, glutamic acid decarboxylase or Zinc transporter 8.
* Patients with known liver disease (other than NAFLD)
* Patients treated with an oral antidiabetic drug, glucagon-like peptide-1 analogues or insulin at the time of or less than 2 weeks prior to inclusion.
* Patients treated with a drug known to affect liver function

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 50 obese children aged 12 to 16 years who have a normal or altered glucose metabolism.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of 1,5-anhydroglucitol levels in obese children with indirect markers of beta-cell function and mass and with metabolic control | First oral glucose tolerance test
  Blood levels of 1,5-anhydroglucitol will be correlated with indirect markers of beta-cell function at 2 timepoints
Correlation of 1,5-anhydroglucitol levels in obese children with indirect markers of beta-cell function and mass and with metabolic control | Second oral glucose tolerance test, 2 years after the first
  Blood levels of 1,5-anhydroglucitol will be correlated with indirect markers of beta-cell function at 2 timepoints

SECONDARY OUTCOMES:
Blood levels of 1,5-anhydroglucitol will be correlated with indicators of the liver function at different moments after diagnosis | First oral glucose tolerance test
  Blood levels of 1,5-anhydroglucitol will be correlated with indicators of the liver function at 2 timepoints
Blood levels of 1,5-anhydroglucitol will be correlated with indicators of the liver function at different moments after diagnosis | Second oral glucose tolerance test, 2 years after the first
  Blood levels of 1,5-anhydroglucitol will be correlated with indicators of the liver function at 2 timepoints

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Geneva, Geneva, Canton of Geneva, Switzerland